CLINICAL TRIAL: NCT00184808
Title: Ambulatory Assessment of Motor State in Patients With Parkinson's Disease in Real Daily Life
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Other Study IDs: dialypd; mar02-0219
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Patients with Parkinson's disease (PD) suffer from motor fluctuations and levodopa induced dyskinesia. The prupose of this study is to evaluate the effect of an automatic system to assess the motor state of PD patients in real daily life. Movements and postures are assessed using 6 accelerometers attached to the the most affected wrist, trunk, both upper legs and both upper arms. Patients wear the system for two days and keep an own diary of their motor state

ELIGIBILITY:
Inclusion Criteria:

Patients with parkinson's disease with motor fluctuations and dyskinesias

Exclusion Criteria:

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15

CONTACTS AND LOCATIONS:
Overall Officials: Stan Gielen, Prof, Study Chair — Radboud University Medical Center; Martin Horstink, MD,PhD, Study Chair — Radboud university Nijmegen medical center
Locations (1):
- Radboud university Nijmegen, Nijmegen, Netherlands